CLINICAL TRIAL: NCT01171846
Title: A Multicentre Randomised Controlled Trial of Pelvic Floor Muscle Training to Prevent Pelvic Organ Prolapse in Women
Brief Title: A Study of the Effects of Physiotherapy to Prevent Pelvic Organ Prolapse
Acronym: PREVPROL
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Glasgow Caledonian University (Other)
Collaborators: University of Birmingham (Other); Birmingham Women's NHS Foundation Trust (Other Government); University of Aberdeen (Other); Aberdeen Royal Infirmary (Other); University of Otago (Other)
Responsible Party: Principal Investigator, Ms Suzanne Hagen, Programme Director, Glasgow Caledonian University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: PREVPROL Study RG1271
Record Dates: First submitted 2010-07-06; First posted 2010-07-29 (Estimated); Last update posted 2015-03-17 (Estimated); Status verified 2015-03

CONDITIONS: Pelvic Organ Prolapse
Keywords: prevention; pelvic floor muscle training; prolapse symptoms; urinary symptoms; sexual function; randomised controlled trial
MeSH Terms: conditions — Pelvic Organ Prolapse

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No

ARMS (2):
- Physiotherapy (Active Comparator)
  Interventions: Other: Pelvic Floor Muscle training
- Control (No Intervention): Women allocated to the Control group will only receive, by post, the same Lifestyle Advice Sheet as the intervention group.

INTERVENTIONS:
Other: Pelvic Floor Muscle training — Women allocated to the intervention group will have five appointments with a specialist women's health physiotherapist (intervention physiotherapist) over 16 weeks who will prescribe a daily exercise programme and provide a Lifestyle Advice Sheet (focusing on weight loss, constipation, avoidance of heavy lifting, coughing and high-impact exercise) and relevant tailored advice (phase 1).
  Thereafter women in the intervention group will be offered Pilates-based classes, including PFMT, as maintenance (phase 2). Classes will be led by a physiotherapist who has undertaken Pilates training and will take place in six week blocks; each woman will be offered two six week blocks over a year. An exercise DVD will be provided for home use. Each woman will be offered a one-to-one review physiotherapy appointment at one and two years after randomisation.
  Arms: Physiotherapy

SUMMARY:
Pelvic organ prolapse is a problem experienced by women where a bulge comes down in the vagina, and may even drop down outside the vagina. The bulge in the vagina is caused by other organs moving down from their normal position in the pelvis and pushing into the vagina. This is a very common problem and many women who have given birth will have a very mild bulge which does not cause them symptoms. Women can however experience a variety of pelvic, bladder, bowel and sexual symptoms which impact on daily life. No research studies have properly examined whether or not exercises can prevent prolapse. This study aims to explore whether exercises taught by a physiotherapist can prevent women developing a prolapse which requires them to have treatment.

ELIGIBILITY:
Inclusion Criteria:

Women involved in the ProLong study who:

* have some evidence of vaginal laxity in any compartment (POP-Q stage I, II or III)
* have had no previous treatment for prolapse (surgery, pessary, PFMT)

Women must be willing to participate in the Trial and to comply with their group allocation.

Exclusion Criteria:

Women:

* with stage 0 or IV prolapse
* who have had previous incontinence surgery (except mid-urethral sling operation)
* who have had previous formal instruction in PFMT for any diagnosis in preceding five years
* who are pregnant, or delivered a baby within the last six months
* who are unable to comply with PFMT treatment
* who are unable to give informed consent

Sex: Female | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 337 (Actual)
Dates: Start 2010-08; Primary Completion 2013-12 (Actual); Study Completion 2013-12 (Actual)

PRIMARY OUTCOMES:
Pelvic organ prolapse symptom score (POP-SS) | Baseline (prior to randomisation)
  A summation of responses to seven prolapse symptom questions (range 0-28)
Pelvic organ prolapse symptom score (POP-SS) | 1 Year post randomisation
  A summation of responses to seven prolapse symptom questions (range 0-28)
Pelvic organ prolapse symptom score (POP-SS) | 2 years post randomisation
  A summation of responses to seven prolapse symptom questions (range 0-28)
Pelvic organ prolapse symptom score (POP-SS) | 3 years post randomisation
  A summation of responses to seven prolapse symptom questions (range 0-28)
Pelvic organ prolapse symptom score (POP-SS) | 4 years post randomisation
  A summation of responses to seven prolapse symptom questions (range 0-28)

SECONDARY OUTCOMES:
Prolapse-related quality of life | Baseline (prior to randomisation)
  Single item scored 0 to 10
Prolapse severity | Four years post randomisation
  Pelvic Organ Prolapse Quantification assessment
Lifestyle changes | 1 year post randomisation
Urinary symptoms | Baseline (prior to randomisation)
  ICIQ urinary incontinence short-form
Bowel symptoms | Baseline (prior to randomisation)
  ICIQ bowel symptoms module
Sexual symptoms | Baseline (prior to randomisation)
  Prolapse Incontinence Sexual Questionnaire - PISQ 12
General health status | Baseline (prior to randomisation)
  SF-12
Need for prolapse treatment | 1 year post randomisation
The average number of days of prolapse symptoms | Baseline (prior to randomisation)
Prolapse-related quality of life | 1 year post randomisation
  Single item scored 0 to 10
Prolapse-related quality of life | 2 years post randomisation
  Single item scored 0 to 10
Prolapse-related quality of life | 3 years post randomisation
  Single item scored 0 to 10
Prolapse-related quality of life | 4 years post of randomisation
  Single item scored 0 to 10
Lifestyle changes | 2 years post randomisation
Lifestyle changes | 3 years post randomisation
Lifestyle changes | 4 years post randomisation
Urinary symptoms | 1 year post randomisation
  ICIQ urinary incontinence short-form
Urinary symptoms | 2 years post randomisation
  ICIQ urinary incontinence short-form
Urinary symptoms | 3 years post randomisation
  ICIQ urinary incontinence short-form
Urinary symptoms | 4 years post randomisation
  ICIQ urinary incontinence short-form
Bowel symptoms | 1 year post randomisation
  ICIQ bowel symptoms module
Bowel symptoms | 2 years post randomisation
  ICIQ bowel symptoms module
Bowel symptoms | 3 years post randomisation
  ICIQ bowel symptoms module
Bowel symptoms | 4 years post randomisation
  ICIQ bowel symptoms module
Sexual symptoms | 1 year post randomisation
  Prolapse Incontinence Sexual Questionnaire - PISQ 12
Sexual symptoms | 2 years post randomisation
  Prolapse Incontinence Sexual Questionnaire - PISQ 12
Sexual symptoms | 3 years post randomisation
  Prolapse Incontinence Sexual Questionnaire - PISQ 12
Sexual symptoms | 4 years post randomisation
  Prolapse Incontinence Sexual Questionnaire - PISQ 12
General health status | 1 year post randomisation
  Prolapse Incontinence Sexual Questionnaire - PISQ 12
General health status | 2 years post randomisation
  Prolapse Incontinence Sexual Questionnaire - PISQ 12
General health status | 3 years post randomisation
  Prolapse Incontinence Sexual Questionnaire - PISQ 12
General health status | 4 years post randomisation
  Prolapse Incontinence Sexual Questionnaire - PISQ 12
Need for prolapse treatment | 2 years post randomisation
Need for prolapse treatment | 3 years post randomisation
Need for prolapse treatment | 4 years post randomisation
The average number of days of prolapse symptoms | 1 year post randomisation
The average number of days of prolapse symptoms | 2 years post randomisation
The average number of days of prolapse symptoms | 3 years post randomisation
The average number of days of prolapse symptoms | 4 years post randomisation

CONTACTS AND LOCATIONS:
Overall Officials: Prof Hagen, PhD MSc BSc CStat CSci, Principal Investigator — NMAHP Research Unit
Locations (3):
- Dunedin School of Medicine, Dunedin, New Zealand
- United Kingdom (2):
  - Aberdeen Royal Infirmary, Aberdeen, Aberdeenshire
  - Birmingham Women's Hospital, Edgbaston, Birmingham

REFERENCES:
- [Result] Hagen, S., C. Glazener, D. McClurg, C. Macarthur, P. Herbison, D. Wilson, P. Toozs-Hobson et al.
- [Derived] Hagen S, Glazener C, McClurg D, Macarthur C, Elders A, Herbison P, Wilson D, Toozs-Hobson P, Hemming C, Hay-Smith J, Collins M, Dickson S, Logan J. Pelvic floor muscle training for secondary prevention of pelvic organ prolapse (PREVPROL): a multicentre randomised controlled trial. Lancet. 2017 Jan 28;389(10067):393-402. doi: 10.1016/S0140-6736(16)32109-2. Epub 2016 Dec 21. PMID 28010994